CLINICAL TRIAL: NCT06536972
Title: Dual-focus Survey with an Emphasis on Heated Humidification Systems
Status: Completed | Type: Observational
Sponsor: Argentinian Intensive Care Society (Other)
Responsible Party: Principal Investigator, Gustavo Plotnikow, Principal investigator, Argentinian Intensive Care Society
Other Study IDs: PRIISABA-CRIHB #12359
Record Dates: First submitted 2024-06-14; First posted 2024-08-05 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-08

CONDITIONS: Survey, Family Life; Knowledge, Attitudes, Practice
Keywords: Heat and moisture exchangers; Heated humidifiers; Questionnaire
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | US Export: No

INTERVENTIONS:
Other: knowledge — Develop an instrument to evaluate knowledge about humidification systems among different health professionals in intensive care units (ICU).
  Describe the knowledge about humidification systems among different health professionals in intensive care units (ICU).

SUMMARY:
Under normal circumstances the upper airway and respiratory tract play a crucial role in humidifying and warming inhaled air, a process known as inspired gas conditioning. This process is essential for effective gas conditioning and mitigating the potential risk of damaging the structure and function of the respiratory epithelium. Airway instrumentation, such as the use of an orotracheal tube or tracheostomy cannula, interferes with the physiological conditioning of inspired gas. Furthermore, the administration of cold, dry medical gases, together with the high flows experienced by patients under invasive mechanical ventilation (IVM) or non-invasive mechanical ventilation (NIMV), exacerbate this unfavorable condition. Therefore, the incorporation of an external device to condition the delivered gas becomes imperative, even in short-term interventions.

There are different devices to condition the inhaled gas, basically passive humidification systems (HMEF) and active (or heated) systems. Considering the humidification capacity and advantages and disadvantages, both passive and active systems are suitable for conditioning the inhaled gas.

The hyphotesis of this study is that health teams in Latin America have limited knowledge regarding humidification systems, both from the technical aspects of implementation and from the clinic.

OBJECTIVES

Primary aim:

Develop an instrument to evaluate knowledge about humidification systems among different health professionals in intensive care units (ICU).

Describe the knowledge about humidification systems among different health professionals in intensive care units (ICU).

Secondary aim:

Compare knowledge about humidification systems between different countries. Compare knowledge about humidification systems between different specialties. Compare knowledge about humidification systems in different age groups.

ELIGIBILITY:
Inclusion Criteria:

* Doctor, nurse, respiratory therapist or related titles
* More than 2 years of work experience in an adult ICU (work in the ICU will be considered as work carried out at least 12 hours per week in the critical care unit)

Exclusion Criteria:

* ≥10% missing survey data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is health professionals who work in Intensive Care Units in Latin America
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Develop questionnaire named "Double-Focus Survey with Emphasis on Active Heated Humidification Systems" | From April 1 to April 30
  Develop an questionnaire to evaluate knowledge about humidification systems among different health professionals in intensive care units (ICU).
Describe the knowledge using the questionnaire previously developed | From June 1 to August 30
  Measure the level of knowledge among different health professionals in ICU settings using the developed questionnaire named "Double-Focus Survey with Emphasis on Active Heated Humidification Systems". This assessment will include evaluating the understanding of the principles, usage, and maintenance of humidification systems.

SECONDARY OUTCOMES:
Compare knowledge about humidification systems between different countries using the questionnaire "Double-Focus Survey with Emphasis on Active Heated Humidification Systems" | From June 1 to August 30
Describe and compare the knowledge about humidification systems between different specialties using the questionnaire "Double-Focus Survey with Emphasis on Active Heated Humidification Systems" | From June 1 to August 30
  Stratification by specialities for describe and compare the knowledge about humidification systems.
Describe and compare knowledge about humidification systems in different age groups using the queationnaire "Double-Focus Survey with Emphasis on Active Heated Humidification Systems" | From June 1 to August 30
  Stratification by age for describe and compare the knowledge about humidification systems.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Britanico de Buenos Aires, Ciudad Autónoma de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] Keck T, Leiacker R, Riechelmann H, Rettinger G. Temperature profile in the nasal cavity. Laryngoscope. 2000 Apr;110(4):651-4. doi: 10.1097/00005537-200004000-00021. PMID 10764013
- [Background] Lindemann J, Leiacker R, Rettinger G, Keck T. Nasal mucosal temperature during respiration. Clin Otolaryngol Allied Sci. 2002 Jun;27(3):135-9. doi: 10.1046/j.1365-2273.2002.00544.x. PMID 12071984
- [Background] Mercke U. The influence of temperature on mucociliary activity. Temperature range 40 degrees C to 50 degrees C. Acta Otolaryngol. 1974 Sep-Oct;78(3-4):253-8. doi: 10.3109/00016487409126352. No abstract available. PMID 4432749
- [Background] Walker AK, Bethune DW. A comparative study of condenser humidifiers. Anaesthesia. 1976 Oct;31(8):1086-93. doi: 10.1111/j.1365-2044.1976.tb11950.x. PMID 1068640
- [Background] Rathgeber J, Kazmaier S, Penack O, Zuchner K. Evaluation of heated humidifiers for use on intubated patients: a comparative study of humidifying efficiency, flow resistance, and alarm functions using a lung model. Intensive Care Med. 2002 Jun;28(6):731-9. doi: 10.1007/s00134-002-1275-9. Epub 2002 Apr 26. PMID 12107679
- [Background] BURTON JD. Effects of dry anaesthetic gases on the respiratory mucous membrane. Lancet. 1962 Feb 3;1(7223):235-8. doi: 10.1016/s0140-6736(62)91187-x. No abstract available. PMID 13875072
- [Background] Dery R. The evolution of heat and moisture in the respiratory tract during anaesthesia with a non-rebreathing system. Can Anaesth Soc J. 1973 May;20(3):296-309. doi: 10.1007/BF03027168. No abstract available. PMID 4704875
- [Background] Eckerbom B, Lindholm CE. Performance evaluation of six heat and moisture exchangers according to the Draft International Standard (ISO/DIS 9360). Acta Anaesthesiol Scand. 1990 Jul;34(5):404-9. doi: 10.1111/j.1399-6576.1990.tb03112.x. PMID 2389657
- [Background] Cohen IL, Weinberg PF, Fein IA, Rowinski GS. Endotracheal tube occlusion associated with the use of heat and moisture exchangers in the intensive care unit. Crit Care Med. 1988 Mar;16(3):277-9. doi: 10.1097/00003246-198803000-00013. PMID 3422625
- [Background] Branson R, Davis K Jr. Evaluation of 21 passive humidifiers according to the ISO 9360 standard: moisture output, dead space, and flow resistance. Respir Care. 1996;41:736-43
- [Background] Unal N, Kanhai JK, Buijk SL, Pompe JC, Holland WP, Gultuna I, Ince C, Saygin B, Bruining HA. A novel method of evaluation of three heat-moisture exchangers in six different ventilator settings. Intensive Care Med. 1998 Feb;24(2):138-46. doi: 10.1007/s001340050535. PMID 9539071
- [Background] Wilkes AR. Heat and moisture exchangers. Structure and function. Respir Care Clin N Am. 1998 Jun;4(2):261-79. PMID 9648186
- [Background] Martin C, Papazian L, Perrin G, Saux P, Gouin F. Preservation of humidity and heat of respiratory gases in patients with a minute ventilation greater than 10 L/min. Crit Care Med. 1994 Nov;22(11):1871-6. PMID 7956294
- [Background] Martin C, Thomachot L, Quinio B, Viviand X, Albanese J. Comparing two heat and moisture exchangers with one vaporizing humidifier in patients with minute ventilation greater than 10 L/min. Chest. 1995 May;107(5):1411-5. doi: 10.1378/chest.107.5.1411. PMID 7750340
- [Background] Plotnikow GA, Accoce M, Navarro E, Tiribelli N. Humidification and heating of inhaled gas in patients with artificial airway. A narrative review. Rev Bras Ter Intensiva. 2018 Mar;30(1):86-97. doi: 10.5935/0103-507x.20180015. PMID 29742220
- [Background] Branson RD. Humidification for patients with artificial airways. Respir Care. 1999;44(6):630-41
- [Background] Oh TE, Lin ES, Bhatt S. Resistance of humidifiers, and inspiratory work imposed by a ventilator-humidifier circuit. Br J Anaesth. 1991 Feb;66(2):258-63. doi: 10.1093/bja/66.2.258. PMID 1817633
- [Background] Roux NG, Plotnikow GA, Villalba DS, Gogniat E, Feld V, Ribero Vairo N, Sartore M, Bosso M, Scapellato JL, Intile D, Planells F, Noval D, Bunirigo P, Jofre R, Diaz Nielsen E. Evaluation of an active humidification system for inspired gas. Clin Exp Otorhinolaryngol. 2015 Mar;8(1):69-75. doi: 10.3342/ceo.2015.8.1.69. Epub 2015 Feb 3. PMID 25729499
- [Background] Ari A, Alwadeai KS, Fink JB. Effects of Heat and Moisture Exchangers and Exhaled Humidity on Aerosol Deposition in a Simulated Ventilator-Dependent Adult Lung Model. Respir Care. 2017 May;62(5):538-543. doi: 10.4187/respcare.05015. Epub 2017 Mar 7. PMID 28270542
- [Background] Thomachot L, Viviand X, Boyadjiev I, Vialet R, Martin C. The combination of a heat and moisture exchanger and a Booster: a clinical and bacteriological evaluation over 96 h. Intensive Care Med. 2002 Feb;28(2):147-53. doi: 10.1007/s00134-001-1193-2. Epub 2002 Jan 12. PMID 11907657
- [Background] Branson RD, Campbell RS, Johannigman JA, Ottaway M, Davis K Jr, Luchette FA, et al. Comparison of conventional heated humidification with a new active hygroscopic heat and moisture exchanger in mechanically ventilated patients. Respir Care. 1999;44(8):912-7.
- [Background] Siempos II, Vardakas KZ, Kopterides P, Falagas ME. Impact of passive humidification on clinical outcomes of mechanically ventilated patients: a meta-analysis of randomized controlled trials. Crit Care Med. 2007 Dec;35(12):2843-51. doi: 10.1097/01.ccm.0000295302.67973.9a. PMID 18074484
- [Background] Kelly M, Gillies D, Todd DA, Lockwood C. Heated humidification versus heat and moisture exchangers for ventilated adults and children. Cochrane Database Syst Rev. 2010 Apr 14;(4):CD004711. doi: 10.1002/14651858.CD004711.pub2. PMID 20393939
- [Background] Klompas M, Branson R, Eichenwald EC, Greene LR, Howell MD, Lee G, Magill SS, Maragakis LL, Priebe GP, Speck K, Yokoe DS, Berenholtz SM. Strategies to prevent ventilator-associated pneumonia in acute care hospitals: 2014 update. Infect Control Hosp Epidemiol. 2014 Sep;35 Suppl 2:S133-54. doi: 10.1017/s0899823x00193894. No abstract available. PMID 25376073
- [Background] Prin S, Chergui K, Augarde R, Page B, Jardin F, Vieillard-Baron A. Ability and safety of a heated humidifier to control hypercapnic acidosis in severe ARDS. Intensive Care Med. 2002 Dec;28(12):1756-60. doi: 10.1007/s00134-002-1520-2. Epub 2002 Oct 8. PMID 12447519
- [Background] American Association for Respiratory Care; Restrepo RD, Walsh BK. Humidification during invasive and noninvasive mechanical ventilation: 2012. Respir Care. 2012 May;57(5):782-8. doi: 10.4187/respcare.01766. PMID 22546299